CLINICAL TRIAL: NCT01001884
Title: The Efficacy of the Caregiver Psychoeducational Consultation Program in Spouse Caregivers of Resectable Colorectal Cancer
Brief Title: The Efficacy of the Caregiver Psychoeducational Consultation Program
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Fei-Hsiu Hsiao, Department of Nursing, College of Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200902029R
Record Dates: First submitted 2009-10-21; First posted 2009-10-27 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-06

CONDITIONS: Depression; Sleep
Keywords: caregiver, psychoeducational, colon
MeSH Terms: conditions — Depression | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- counseling (Experimental): caregiver psychoeducational consultation program (CPCP)
  Interventions: Other: caregiver psychoeducational consultation program (CPCP)

INTERVENTIONS:
Other: caregiver psychoeducational consultation program (CPCP) — 6-session caregiver psychoeducational consultation program (CPCP)
  Other Names: consultation

SUMMARY:
Aim:

To examine the effects of the caregiver psychoeducational consultation program in reducing caregiver burdens, depression, sleep quality, and improving the experience in close relationship, positive meaning of illness and quality of life.

This is the 2-year study. The design adopts the randomized controlled trial (RCT). The caregivers of patients with spouse caregivers of resectable metastatic colorectal cancer will be randomly assigned into two groups: one group receiving usual care, another group receiving the caregiver psychoeducational consultation program (CPCP). The usual care includes providing education materials only. Measurement time-points include pre intervention, post intervention, & then 1, and 3 months after the end of intervention for the maintenance effect.

DETAILED DESCRIPTION:
To examine the effects of the caregiver psychoeducational consultation program in reducing caregiver burdens, depression, sleep quality, and improving the experience in close relationship, positive meaning of illness and quality of life.

This is the 2-year study. The design adopts the randomized controlled trial (RCT). The caregivers of patients with spouse caregivers of resectable metastatic colorectal cancer will be randomly assigned into two groups: one group receiving usual care, another group receiving the caregiver psychoeducational consultation program (CPCP). The usual care includes providing education materials only. Measurement time-points include pre intervention, post intervention, & then 1, and 3 months after the end of intervention for the maintenance effect.

ELIGIBILITY:
Inclusion Criteria:

* Spouse caregivers of patients with resectable colorectal cancer,
* Those who are willing to participate in the research,
* Aged above 18.

Exclusion Criteria:

* Who refuses to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Short-form 12 health-related quality of life questionnaire | pre intervention, post intervention, 1, and 3,months after the end of the interventions

SECONDARY OUTCOMES:
Caregiver reaction assessment | pre intervention, post intervention, 1, and 3,months after the end of the interventions
Experiences in close relationships scale | pre intervention, post intervention, 1, and 3,months after the end of the interventions
Moss sleeping scale | pre intervention, post intervention, 1, and 3,months after the end of the interventions
BDI-II depression scale | pre intervention, post intervention, 1, and 3,months after the end of the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Fei Hsiao, PhD, Principal Investigator — Department of Nursing, College of Medicine, National Taiwan University
Locations (1):
- Fei-Hsiu Hsiao, Taipei, Taiwan